CLINICAL TRIAL: NCT05314088
Title: Testing the Efficacy and Mechanisms of an Adapted Resilience Building Intervention in People Aging With HIV
Acronym: RISE+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Pariya L. Fazeli, PhD, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB-300008740; 1R21AG076377-01A1 (NIH)
Record Dates: First submitted 2022-03-21; First posted 2022-04-06 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Resilience; HIV-1-infection; Stress, Psychological
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: A two group RCT, one group receives the behavioral intervention and one receives an attention matched placebo control intervention.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RISE+ Resilience Intervention (Experimental): Participants in the intervention group will come to the lab for four two-hour weekly sessions in small groups of 3-4. The intervention includes psychoeducational videos and individual written activities on topics such as coping strategies, cognitive appraisals, the responsibility model, and social connections, all integrated into the overarching process of resilience. The intervention will be facilitated by a trained research assistant but as in the pilot study, he/she will be minimally involved (i.e., only administering the videos and explaining the activities) to keep the private reflective nature of the program that participants liked. Upon completion of the program, participants will be given handouts with summaries of the program material. We will gather qualitative and quantitative feedback on the intervention at the one-month posttest.
  Interventions: Behavioral: RISE+
- Stress Reduction Control (Placebo Comparator): Control participants will complete an attention-matched internet stress reduction paradigm, which includes an internet navigation protocol and placebo computer games. As with the intervention group, participants in the control group will come to the lab for four two-hour weekly sessions in small groups of 3-4. Facilitator involvement will be the same as the intervention group (e.g., the research assistant will explain computer activities and games but will otherwise not interact with the participant).
  Interventions: Behavioral: Stress Reduction Control

INTERVENTIONS:
Behavioral: RISE+ — The intervention includes psychoeducational videos and written activities on topics such as coping strategies, cognitive appraisals, the responsibility model, and social connections, all integrated into the overarching process of resilience.
  Arms: RISE+ Resilience Intervention
Behavioral: Stress Reduction Control — Placebo Comparator: Stress Reduction Control Control participants will complete an attention-matched internet stress reduction paradigm, which includes an internet navigation protocol and placebo computer games.
  Arms: Stress Reduction Control

SUMMARY:
This study will examine the mechanisms and efficacy of a resilience building intervention in older people living with HIV.

DETAILED DESCRIPTION:
A two-group RCT will enroll 100 older (aged 50+) people living with HIV (PLHIV), who will be recruited from the UAB HIV outpatient clinic. Eligible participants will complete a baseline assessment including a 14-day experience sampling method (ESM) protocol, and then be randomized to either the intervention group (n=50) or an attention-matched control group (n=50). We will block randomize groups based on race, sex, and self-reported resilience (Connor Davidson Resilience Scale). If differences are found between groups on influential variables (e.g., SES), such factors will be controlled in analyses and exploratory aim analyses will examine treatment moderators (e.g., sex, race). Both groups will return for four weekly two-hour group visits, followed by a one-month post intervention assessment (including qualitative and quantitative feedback) and a second ESM protocol. A three-month follow-up (comparable to baseline) will assess health outcomes. A blinded research assistant will conduct follow-ups. Our Primary Aims will use ESM via text messaging, and focus on intervention effects on the use of resilience resources following times when stressors are reported and whether such increases drive improved affective stress reactivity and recovery (Aim 1). Our secondary aim will examine effects on health outcomes at three months. Our exploratory aim will examine moderators of treatment response.

ELIGIBILITY:
Inclusion Criteria:

* current UAB HIV Clinic patient
* age 50+
* have a recent history (within the past 12 months) of suboptimal HIV management, defined as having either ≥one record of detectable viral load or ≥one missed clinic visit without prior cancellation/reschedule

Exclusion Criteria:

* neurological or severe psychiatric (e.g., schizophrenia, bipolar disorder, major depression) disorders

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
resilience resources | immediately following the 4 week intervention
  we will use daily text messaging after the intervention to assess use of resilience resources following stressors. Participants will be texted daily to ask if they experienced a stressor (YES/NO) and then they respond on a 5 pt Likert scale on their levels of 7 resilience resources: hardiness, optimism, self-efficacy, locus of control, positive reframing, proactive coping, and social support. Scores will be a total average score and individual average scores for each resource.
stress reactivity | immediately following the 4 week intervention
  we will use daily text messaging after the intervention to assess use of stress reactivity following stressors. Participants will be texted daily to ask if they experienced a stressor (YES/NO) and then they respond on a Visual Analog Scale of their positive and negative affect. Their are 10 items for positive affect and 10 for negative affect. Total average positive and negative affect scores will be used.

SECONDARY OUTCOMES:
health related quality of life | 3 months after intervention
  Medical Outcomes Study HIV Health Survey
depressive symptoms | 3 months after intervention
  Centers for Epidemiological Studies Depression Scale
HIV medication adherence | 3 months after intervention
  Visual Analogue Scale ART adherence
HIV Treatment Management Abilities | 3 months after intervention
  HIV Treatment Adherence Self-Efficacy Scale
HIV Viral Load | 3 months after intervention
  HIV plasma viral load (copies per mL of plasma) extracted from medical records

CONTACTS AND LOCATIONS:
Locations (1):
- Holley Mears Building, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No